CLINICAL TRIAL: NCT04929990
Title: The Therapeutic Effect of Inspiratory and Expiratory Muscle Strengthening Training on Patients With COPD and Mild Cognitive Impairment
Brief Title: The Effect of Respiratory Muscle Training for Patients With COPD and Mild Cognitive Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CF18259A
Record Dates: First submitted 2021-06-03; First posted 2021-06-18 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Chronic Obstructive Pulmonary Disease; Mild Cognitive Impairment
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Cognitive Dysfunction | interventions — Breathing Exercises

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inpiratory and expiratory muscle training (Experimental): The initial intensity of training was set on 30% of the MIP and MEP for inspiratory and expiratory muscle training, respectively. The intensity was adjusted to add 5% of resistance each week
  Interventions: Behavioral: Respiratory muscle training
- Inspiratory muscle training (Active Comparator): The initial resistance of the breathing trainer was also set on 30% of MIP, and the following adjustments were also in accordance to the protocol of the experimental group
  Interventions: Behavioral: Respiratory muscle training

INTERVENTIONS:
Behavioral: Respiratory muscle training — Inspiratory and expiratory muscle training were performed using a breathing trainer (Dofin DT11/14, Galemed Co. Ltd, Taiwan) for 30 minutes a day with a total of eight weeks. Before the training, the MIP and maximal expiratory pressure (MEP) were documented by the best performance of three trials with a digital pressure gauge (GB60, Jitto International Co. Ltd, Taiwan)

SUMMARY:
Patients with COPD and MCI received either inspiratory muscle training or inspiratory plus expiratory muscle training and compared the therapeutic effects

DETAILED DESCRIPTION:
Patients with COPD and MCI were recruited, and were randomly assigned to the experimental group and the control group. The experimental group consisted of EMT and IMT for a total of 8 weeks, while the control group received IMT only. Outcomes measured and compared in this cohort were diaphragmatic thickness fraction and excursion examined by ultrasound, the dyspnea score of modified Medical Research Council (mMRC), the cognitive score of Mini-Mental State Examination (MMSE), and the score of COPD Assessment Test (CAT). In addition, the pulmonary function test, the cardiopulmonary exercise test, and the physiology performance of six minute walking test were also obtained. We also analyzed the difference of each parameters before and after training in each patient.

ELIGIBILITY:
Inclusion Criteria:

* 1. Having definite diagnosis of COPD, namely the value of the FEV1 divided by forced vital capacity (FVC) 10 to 15 minutes after beta-2 agonist inhalation being less than 0.7.
* 2. The score of Mini-Mental State Examination (MMSE) being between 23 and 27

Exclusion Criteria:

* 1. Being not able to follow instructions on respiratory muscle training or complete the questionnaires of our study due to cognitive impairment.
* 2. Having difficulty to complete the cardiopulmonary exercise testing or the six minute walking test (6MWT) due to high risk cardiopulmonary diseases or other orthopedic conditions.
* 3. Having the diagnosis of lung cancer or history of receiving thoracoabdominal surgery
* 4. Having Body Mass Index more than 30

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2018-08-07 (Actual); Primary Completion 2021-04-06 (Actual); Study Completion 2021-06-02 (Actual)

PRIMARY OUTCOMES:
MMSE | 8 weeks
  Mini-Mental State Examination

SECONDARY OUTCOMES:
Diaphragmatic thickness fraction | 8 weeks
  Diaphragmatic thickness fraction on ultrasonography
chronic obstructive pulmonary disease assessment test (CAT) | 8 weeks
  questionnaire of dyspnea
diffusing capacity of the lung for carbon monoxide (DLCO) | 8 weeks
  diffusing capacity of the lung for carbon monoxide (DLCO) in pulmonary function test
dead space fraction (Vd/Vt) | 8 weeks
  dead space fraction (Vd/Vt) in cardiopulmonary function test
the distance walked in 6 minutes | 8 weeks
  the distance walked in 6 minutes
Diaphragmatic excursion | 8 weeks
  Diaphragmatic excursion on ultrasonography
forced vital capacity | 8 weeks
  forced vital capacity tested in pulmonary function test
forced expiratory volume in 1 second | 8 weeks
  forced expiratory volume in 1 second in pulmonary function test
forced expiratory volume in 1 second divided by forced vital capacity | 8 weeks
  forced expiratory volume in 1 second divided by forced vital capacity in pulmonary function test
DLCO divided by alveolar volume (VA) | 8 weeks
  DLCO divided by alveolar volume (VA) in pulmonary function test
modified Medical Research Council (mMRC) | 8 weeks
  questionnaire of dyspnea
minute ventilation to carbon dioxide output (VE/VCO2) slope | 8 weeks
  minute ventilation to carbon dioxide output (VE/VCO2) slope in cardiopulmonary function test
the change of oxygen saturation in 6 minutes walking test | 8 weeks
  the change of oxygen saturation in 6 minutes walking test
the change of Borg scale in 6 minutes walking test | 8 weeks
  the change of Borg scale in 6 minutes walking test

CONTACTS AND LOCATIONS:
Overall Officials: Yuan-Yang Cheng, Study Director — Taichung Veterans General Hospital
Locations (1):
- Taichung Veterans General Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No